CLINICAL TRIAL: NCT03886597
Title: Table Olives Nutritional Intervention: Pharmacokinetics of Polyphenols and Pentacyclic Triterpenes and Assessment of Antioxidant, Cardiovascular and Anti-inflammatory Biomarkers
Brief Title: Nutritional Intervention With Table Olives in Healthy Volunteers
Acronym: BIOLIVA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Ministerio de Economía y Competitividad (Spain) AGL 2013-41188R (Unknown); University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IIBSP-OLI-2016-23
Record Dates: First submitted 2019-03-15; First posted 2019-03-22 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Healthy; Biological Availability; Nutritional Intervention; Functional Food; Nutrition Physiology
Keywords: Polyphenols; Triterpenes; Olea europaea; Table Olives; Pharmacokinetics; Functional Food; Antioxidant; Cardiovascular Disease; Anti-inflammatory
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This study involve two stages, the first one corresponding to the pharmacokinetic study of the single administration of table olives in healthy male volunteers and the second one corresponding to the study of a nutritional intervention with 30 table olives during 30 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 60 Arbequina Table Olives (Experimental): Pharmacokinetics Study
  Interventions: Other: Table Olives
- 120 Arbequina Table Olives (Experimental): Pharmacokinetics Study
  Interventions: Other: Table Olives
- 60 Table Olives (Experimental): Table Olives Nutritional Intervention
  Interventions: Other: Table Olives
- Control (No Intervention): Control of Table Olives Nutritional Intervention

INTERVENTIONS:
Other: Table Olives — At early morning (08:00 h e.g.) and after 10 hours of fasting conditions, the olives of the Arbequina variety will be administered to each subject. The 60 olives will be weighted before the ingestion and the remaining stones will be subsequently weighted to keep a record of the amount of olive pulp that has been consumed. The subjects will have a period of 5 minutes to ingest 60 olives with 240 mL of water. Blood samples will be collected from 1 hour prior to administration until 24 hours after dosing. Urine samples will also be collected and blood pressure will be measured.
  Arms: 60 Arbequina Table Olives
Other: Table Olives — At early morning (08:00 h e.g.) and after 10 hours of fasting conditions, the olives of the Arbequina variety will be administered to each subject. The 120 olives will be weighted before the ingestion and the remaining stones will be subsequently weighted to keep a record of the amount of olive pulp that has been consumed. The subjects will have a period of 10 minutes to ingest 120 olives with 240 mL of water. Blood samples will be collected from 1 hour prior to administration until 24 hours after dosing. Urine samples will also be collected and blood pressure will be measured.
  Arms: 120 Arbequina Table Olives
Other: Table Olives — All the subjects will perform two experimental sessions of 30 days with 15 days of washout periods within experimental periods. In one experimental session subjects will ingest table olives and in the other session they will act as their own controls following their normal dietary habits. During all the experiment participants will avoid the consumption of products rich in phenolic and triterpenic compounds. Subjects will include the dose of 60 table olives within their normal dietary habits. Consequently, the olives will be consumed two times daily within each main meal; 30 olives before lunch and 30 olives before dinner. Blood samples will be collected at baseline and 15 and 30 days of each experimental session. Tolerability variables and blood pressure will also be measured.
  Arms: 60 Table Olives

SUMMARY:
Olives and olive oil are typical components of the Mediterranean diet being part of its cultural and gastronomic heritage. Since ancient times, olives have been used either for both, oil extraction or whole fruit consumption as table olives. Olive oil stands out from both the nutritional and the health point of view. However, the effect of table olives consumption remains almost unknown. The beneficial properties of olive oil have been initially ascribed to the high concentration of oleic acid. Nowadays, these positive effects have been attributed also to minor compounds such as polyphenols or pentacyclic triterpenes. Table olives contain a higher amount of both polyphenols and pentacyclic triterpenes than their oil, with the same healthy fatty acid profile. Therefore, the present intervention aims at investigating the pharmacokinetic of polyphenols and pentacyclic triterpenes after a single olive intake as well as the assessment of the effect of the consumption of olives during 30 days on the overall health status playing particular attention to the anti-inflammatory, antioxidant and cardiovascular biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 19 and 30 kg/m2.
* Healthy on the basis of physical examination and routine biochemical and hematological laboratory determinations.
* Free acceptance to participate in the study by obtains signed informed consent.

Exclusion Criteria:

* Smoking.
* Alcohol or drug abuse.
* Heavy consumer of stimulating beverages (>5 coffees, teas, chocolate or cola drinks per day) and grapefruit juice.
* Background of allergy, idiosyncrasy or hypersensitivity to drugs.
* Intake of any medication within 2 weeks prior taking the study intervention (except for use of paracetamol in short-term symptomatic treatments), including over-the-counter products (including natural food supplements, vitamins and medicinal plants products), or any enzymatic inductor or inhibitor within 3 months before the drug administration.
* Positive serology for hepatitis B, C or HIV.
* Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological or neurological disease or other chronic diseases.
* Having undergone major surgery during the previous 6 months.
* Pregnancy or lactation status (if applied).
* Participation in another clinical trial during the 3 months preceding the drug administration.
* Donation of blood during the 4 weeks preceding the drug administration.
* Acute illness four weeks before drug administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Stage 1: Maximum plasma concentration (Cmax) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Concentration at the end of the dosing interval (Ct) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Time until Cmax is reached (Tmax) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Area under the curve from administration to last observed concentration at time (AUC (0-t) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: AUC extrapolated to infinite time (AUC (0-∞) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Percentage of AUC extrapolated (AUC%) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Terminal elimination rate constant (Kel) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Plasma concentration half-life (t ½) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Volume of distribution (Vd/ F) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Clearance (Cl/F) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Peak trough fluctuation over one dosing interval at steady state (PTF) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Cmax dose normalized (Cmax/Dose) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: AUC (0-t) dose normalized (AUC (0-t)/Dose) | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Urine polyphenols concentration | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 1: Urine triterpenes concentration | 24 hours
  24 hour dosing period; 2 dosing periods each separated by 7 days washout
Stage 2: Plasma polyphenols concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Plasma triterpenes concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Urine polyphenols concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Urine triterpenes concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Malondialdehyde concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Catalase concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Glutathione peroxidase concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Superoxide dismutase concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: F2A isoprostane concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: 8 isoprostane concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Oxidized low-density lipoprotein concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: C-Reactive Protein concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Lipoprotein-associated phospholipase A2 concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Apolipoprotein A1 concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Apolipoprotein B100 concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Tumor necrosis factor alpha concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Interleukin 6 concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Interleukin 1 concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days

SECONDARY OUTCOMES:
Stage 1 and 2: Number of participants with treatment-related adverse events | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 1 and 2: Systolic and diastolic blood pressure | Stage 1: 24 hour dosing period; 2 dosing periods each separated by 7 days washout, Stage 2: 30 days dosing period or 30 days as control group separated by 15 days washout
  Stage 1: 24 hours, Stage 2: 30 days
Stage 1 and 2: Heart rate | Stage 1: 24 hour dosing period; 2 dosing periods each separated by 7 days washout, Stage 2: 30 days dosing period or 30 days as control group separated by 15 days washout
  Stage 1: 24 hours, Stage 2: 30 days
Stage 1 and 2: Respiratory rate | Stage 1: 24 hour dosing period; 2 dosing periods each separated by 7 days washout, Stage 2: 30 days dosing period or 30 days as control group separated by 15 days washout
  Stage 1: 24 hours, Stage 2: 30 days
Stage 2: Body weight | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: High-density lipoprotein cholesterol concentration (HDL-C) | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Low-density lipoprotein cholesterol concentration (LDL-C) | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Very low-density lipoprotein cholesterol concentration (VLDL-C) | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Triglyceride concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Total cholesterol concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Sodium concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Glucose concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Urea concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Creatinine concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Aspartate aminotransferase concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Alanine aminotransferase concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Alkaline phosphatase concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days
Stage 2: Total proteins concentration | 30 days dosing period or 30 days as control group separated by 15 days washout
  30 days

CONTACTS AND LOCATIONS:
Overall Officials: Joana M Planas, PhD Prof., Study Director — Departament de Bioquímica i Fisiologia. Facultat de Farmàcia i Ciències de l´Alimentació. Universitat de Barcelona
Locations (1):
- Institut de Recerca Hospital de la Santa Creu i Sant Pau - CIM Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bachhav SS, Bhutada MS, Patil SP, Sharma KS, Patil SD. Oleanolic Acid Prevents Increase in Blood Pressure and Nephrotoxicity in Nitric Oxide Dependent Type of Hypertension in Rats. Pharmacognosy Res. 2014 Oct-Dec;7(4):385-92. doi: 10.4103/0974-8490.159575. PMID 26692754
- [Background] Cicerale S, Conlan XA, Sinclair AJ, Keast RS. Chemistry and health of olive oil phenolics. Crit Rev Food Sci Nutr. 2009 Mar;49(3):218-36. doi: 10.1080/10408390701856223. PMID 19093267
- [Background] Covas MI, Nyyssonen K, Poulsen HE, Kaikkonen J, Zunft HJ, Kiesewetter H, Gaddi A, de la Torre R, Mursu J, Baumler H, Nascetti S, Salonen JT, Fito M, Virtanen J, Marrugat J; EUROLIVE Study Group. The effect of polyphenols in olive oil on heart disease risk factors: a randomized trial. Ann Intern Med. 2006 Sep 5;145(5):333-41. doi: 10.7326/0003-4819-145-5-200609050-00006. PMID 16954359
- [Background] de la Torre-Carbot K, Chavez-Servin JL, Jauregui O, Castellote AI, Lamuela-Raventos RM, Fito M, Covas MI, Munoz-Aguayo D, Lopez-Sabater MC. Presence of virgin olive oil phenolic metabolites in human low density lipoprotein fraction: determination by high-performance liquid chromatography-electrospray ionization tandem mass spectrometry. Anal Chim Acta. 2007 Feb 5;583(2):402-10. doi: 10.1016/j.aca.2006.10.029. Epub 2006 Nov 2. PMID 17386573
- [Background] Dzubak P, Hajduch M, Vydra D, Hustova A, Kvasnica M, Biedermann D, Markova L, Urban M, Sarek J. Pharmacological activities of natural triterpenoids and their therapeutic implications. Nat Prod Rep. 2006 Jun;23(3):394-411. doi: 10.1039/b515312n. Epub 2006 May 3. No abstract available. PMID 16741586
- [Background] Ghanbari R, Anwar F, Alkharfy KM, Gilani AH, Saari N. Valuable nutrients and functional bioactives in different parts of olive (Olea europaea L.)-a review. Int J Mol Sci. 2012;13(3):3291-3340. doi: 10.3390/ijms13033291. Epub 2012 Mar 12. PMID 22489153
- [Background] Juan ME, Planas JM, Ruiz-Gutierrez V, Daniel H, Wenzel U. Antiproliferative and apoptosis-inducing effects of maslinic and oleanolic acids, two pentacyclic triterpenes from olives, on HT-29 colon cancer cells. Br J Nutr. 2008 Jul;100(1):36-43. doi: 10.1017/S0007114508882979. Epub 2008 Feb 26. PMID 18298868
- [Background] Kountouri AM, Mylona A, Kaliora AC, Andrikopoulos NK. Bioavailability of the phenolic compounds of the fruits (drupes) of Olea europaea (olives): impact on plasma antioxidant status in humans. Phytomedicine. 2007 Oct;14(10):659-67. doi: 10.1016/j.phymed.2007.06.001. Epub 2007 Sep 17. PMID 17870451
- [Background] Liu J, Sun H, Duan W, Mu D, Zhang L. Maslinic acid reduces blood glucose in KK-Ay mice. Biol Pharm Bull. 2007 Nov;30(11):2075-8. doi: 10.1248/bpb.30.2075. PMID 17978478
- [Background] Lou-Bonafonte JM, Arnal C, Navarro MA, Osada J. Efficacy of bioactive compounds from extra virgin olive oil to modulate atherosclerosis development. Mol Nutr Food Res. 2012 Jul;56(7):1043-57. doi: 10.1002/mnfr.201100668. PMID 22760979
- [Background] Lozano-Mena G, Sanchez-Gonzalez M, Juan ME, Planas JM. Maslinic acid, a natural phytoalexin-type triterpene from olives--a promising nutraceutical? Molecules. 2014 Aug 4;19(8):11538-59. doi: 10.3390/molecules190811538. PMID 25093990
- [Background] Madlala HP, Van Heerden FR, Mubagwa K, Musabayane CT. Changes in Renal Function and Oxidative Status Associated with the Hypotensive Effects of Oleanolic Acid and Related Synthetic Derivatives in Experimental Animals. PLoS One. 2015 Jun 5;10(6):e0128192. doi: 10.1371/journal.pone.0128192. eCollection 2015. PMID 26046776
- [Background] Marrugat J, Covas MI, Fito M, Schroder H, Miro-Casas E, Gimeno E, Lopez-Sabater MC, de la Torre R, Farre M; SOLOS Investigators. Effects of differing phenolic content in dietary olive oils on lipids and LDL oxidation--a randomized controlled trial. Eur J Nutr. 2004 Jun;43(3):140-7. doi: 10.1007/s00394-004-0452-8. Epub 2004 Jan 6. PMID 15168036
- [Background] Martin-Pelaez S, Covas MI, Fito M, Kusar A, Pravst I. Health effects of olive oil polyphenols: recent advances and possibilities for the use of health claims. Mol Nutr Food Res. 2013 May;57(5):760-71. doi: 10.1002/mnfr.201200421. Epub 2013 Mar 1. PMID 23450515
- [Background] Melliou E, Zweigenbaum JA, Mitchell AE. Ultrahigh-pressure liquid chromatography triple-quadrupole tandem mass spectrometry quantitation of polyphenols and secoiridoids in california-style black ripe olives and dry salt-cured olives. J Agric Food Chem. 2015 Mar 11;63(9):2400-5. doi: 10.1021/jf506367e. Epub 2015 Feb 26. PMID 25668132
- [Background] Poudyal H, Campbell F, Brown L. Olive leaf extract attenuates cardiac, hepatic, and metabolic changes in high carbohydrate-, high fat-fed rats. J Nutr. 2010 May;140(5):946-53. doi: 10.3945/jn.109.117812. Epub 2010 Mar 24. PMID 20335636
- [Background] Rodriguez-Rodriguez R, Perona JS, Herrera MD, Ruiz-Gutierrez V. Triterpenic compounds from "orujo" olive oil elicit vasorelaxation in aorta from spontaneously hypertensive rats. J Agric Food Chem. 2006 Mar 22;54(6):2096-102. doi: 10.1021/jf0528512. PMID 16536581
- [Background] Sanchez-Quesada C, Lopez-Biedma A, Warleta F, Campos M, Beltran G, Gaforio JJ. Bioactive properties of the main triterpenes found in olives, virgin olive oil, and leaves of Olea europaea. J Agric Food Chem. 2013 Dec 18;61(50):12173-82. doi: 10.1021/jf403154e. Epub 2013 Nov 22. PMID 24279741
- [Background] Uylaser V, Yildiz G. The historical development and nutritional importance of olive and olive oil constituted an important part of the Mediterranean diet. Crit Rev Food Sci Nutr. 2014;54(8):1092-101. doi: 10.1080/10408398.2011.626874. PMID 24499124
- [Background] Weinbrenner T, Fito M, de la Torre R, Saez GT, Rijken P, Tormos C, Coolen S, Albaladejo MF, Abanades S, Schroder H, Marrugat J, Covas MI. Olive oils high in phenolic compounds modulate oxidative/antioxidative status in men. J Nutr. 2004 Sep;134(9):2314-21. doi: 10.1093/jn/134.9.2314. PMID 15333722